CLINICAL TRIAL: NCT04208906
Title: Validation of Masimo O3 Regional Oximetry Device in Pediatric Patients Undergoing Cardiac Surgery
Brief Title: Masimo O3 Regional Oximetry Device in Pediatric Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H1911-099-1081
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Pediatric Cardiac Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with congenital cardiac disease (Experimental): Pediatric patients aged < 7 years undergoing cardiac surgery
  Interventions: Device: Masimo O3

INTERVENTIONS:
Device: Masimo O3 — After anesthesia induction, a masimo O3 sensors are attached to the forehead (ScO2) and the sole of the foot (StO2). About 0.4 ml blood samples are obtained from arterial line and central venous line at three epochs before and after cardiopulmonary bypass (total 6 times)
  * T1: before cardiopulmonary bypass (CPB), fraction of inspired oxygen (FiO2) 0.2
  * T2: before CPB, FiO2 0.5
  * T3: before CPB, FiO2 0.8
  * T4: after CPB, FiO2 0.8
  * T5: after CPB, FiO2 0.5
  * T6: after CPB, FiO2 0.2
  Hemoglobin oxygen saturation values are confirmed in each sample (arterial sample: SaO2, venous sample: SvO2). Each O3 values (ScO2 and StO2) are compared to the values of SvO2, 0.7 × SvO2 + 0.3 × SaO2.

SUMMARY:
We evaluate the relationship between the regional tissue oxygenation value (ScO2 - cerebral, StO2 - lower limb) and mixed venous saturation (SvO2) and arterial oxygen saturation (SaO2) measured before and after correction surgery in pediatric patients undergoing cardiac surgery.

In addition, we compared the sCO2 and sTO2 with reference value which is calculated using SvO2 and SaO2.

ELIGIBILITY:
Inclusion Criteria:

* children under 7 years old

Exclusion Criteria:

* Hyperbilirubinemia
* Skin disease at sensor attachment site
* Single ventricle physiology

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Validation of Masimo O3 value | During surgery
  Comparison of ScO2 and StO2 to reference level (SvO2, 0.7×SvO2 + 0.3×SaO2)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Other, South Korea

REFERENCES:
- [Derived] Lee JH, Song IS, Kang P, Ji SH, Jang YE, Kim EH, Kim HS, Kim JT. Validation of the Masimo O3 regional oximetry device in pediatric patients undergoing cardiac surgery. J Clin Monit Comput. 2022 Dec;36(6):1703-1709. doi: 10.1007/s10877-022-00815-3. Epub 2022 Feb 15. PMID 35169968